CLINICAL TRIAL: NCT03475095
Title: A Mechanism of Tuina Treating Lumbar Disc Herniation Based of Central Nervous System Motion Control Modulating Reconstruction of Lumbar Stabilizer Function
Brief Title: Motor Control Mechanisms by CNS of Tuina in Patients With Lumbar Disk Herniation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LDH-001
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Low Back Pain; Disc, Herniated
Keywords: Low Back Pain; Tuina therapy; lumbar disc herniation; central motion control; functional magnetic resonanceimaging; effect mechanism; Chronic nonspecific low Back pain
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDH patients (Experimental): "ribs and bones" Tuina therapy According to the diagnostic criteria of"vertebral dislocation",determine the position,degree and direction of the dislocation,assess the activity of the affected vertebrae.Treated with combining Tuina of muscle-loosing and bone-setting such as reinforcing ribs，kneading and plucking method,20 min every treatment,twice a week for a total time of 4 weeks.
  Interventions: Other: Tuina

INTERVENTIONS:
Other: Tuina — Patients will receive Tuina therapies tiwce per week in one month.each time lasts about 20 minutes,a total of 4 weeks.

SUMMARY:
Lumbar disk herniation (LDH)is a prevalent health problem around the world. It can cause symptoms of low back pain, numbness or weakness.The understanding of low back pain in traditional Chinese medicine(TCM) theory"unbalanced bones and muscles"that is consistent with the description of modern medicine on LDH function pathology. Tuina is one of Diagnosis and treatment methods in TCM which has been used as a noninvasive treatment of LDH. However, the mechanism of Tuina therapy in LDH is still unclear.The purpose of this study is to establish a platform of the therapeutic effect and mechanical effect of LDH in the treatment of LDH，explore the characteristics of Tuina by the motor control in lumbar CNS,observe the patterns and regularities in the function of related brain regionin of patients with acute or chronic LDH and reveal the mechanism of Tuina of improving the control of lumbar spine CNS movement.

DETAILED DESCRIPTION:
Clinical researches has demonstrated the effectiveness of Tuina on lumbar disc herniation (LDH), but the mechanism remains unclear.The existing researches mainly focus on the mechanical mechanism of the local stability reconstruction of the lumbar spine. Our previous study found that LDH patients have lumbar CNS motion control disorder, and preliminary studies have shown that Tuina can improve the lumbar CNS motion control efficiency, also fMRI studies found that abnormal motion related brain areas had an active trend during the acute phase and a suppressed trend in the chronic period.Therefore,we hypothesize that Tuina could improve the lumbar CNS motion control in LDH patients, and could response to the effect of local mechanical lumbar as well as bidirectionally regulate the function of lumbar stabilizers, which facilitates the stable reconstruction of lumbar. This project will illuminate the effect of Tuina improving the lumbar CNS motion control by applying the latest fMRI, surface electromyography and data mining technology to the acute and chronic LDH patients with a combination of efficacy and experimental verification to reveal the mechanism of CNS bidirectional regulation of paraspinal muscle activity by the response of related brain regions to mechanical effects after Tuina on the lumbar. This project provides a new thinking to the research of the therapeutic mechanism of LDH, which is a scientific significance.

ELIGIBILITY:
Inclusion Criteria:

* accord with the diagnostic criteria of lumbar disc herniation in the seventh edition of "Surgery", and diagnosed by MRI, the course of acute patients ≤ 1 month, the course of chronic patients ≥ 3 months
* Age:25～40 years old
* VAS score ≥30/100
* Waist ODI index≥20%
* Self-rating anxiety scale (SAS)<59 points, Self-rating Depression Scale (SDS) <53 points
* BMI<24
* Signed the Informed Consent Form

Exclusion Criteria:

* History of spinal surgery or history of severe spine trauma
* Combined with other lumbar conditions may interfere with clinical outcomes (e.g. bone tuberculosis, tumors and severe osteoporosis)
* Combines cardiovascular disease, blood system, digestive system and other serious medical diseases or psychosis
* Women at childbearing age and of pregnancy desire during the study
* combined with autoimmune diseases, allergy Sexual diseases, acute and chronic infectious diseases
* Presence of any major physical or neurological illness
* MRI contraindication
* MRI showed nucleus pulposus free, cauda equina syndrome
* vision loss, vestibular dysfunction

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-10 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale (VAS) | 6 weeks
  Assessment of pain intensity before treatment of all patients,collate related data and statistically analyzed.
Oswestry Disability Index (ODI) | 6 weeks
  Assessment of symptoms and severity of low back pain
Biering-Sørensen test | 6 weeks
  Assessment of endurance of the lumbar paraspinal muscle
Rapid reaction time | 6 weeks
  Measurement of rapid reaction time will be conducted in surface electromyo gram

SECONDARY OUTCOMES:
Finite element analysis | 12 weeks
  Intervertebral disc biomechanical analysis
Resting state functional magnetic resonance imaging and magnetic resonance spectroscopy | 12 weeks
  Identification of brain activation in the motor area during Tuina.
Visual analogue scale (VAS) | 12 weeks
  Assessment of pain intensity before treatment of all patients,collate related
Oswestry Disability Index (ODI) | 12 weeks
  Assessment of symptoms and severity of low back pain
Biering-Sørensen test | 12 weeks
  Assessment of endurance of the lumbar paraspinal muscle
Cross sectional area of multifidus | 12 weeks
  Measurement of Cross Sectional Area of Multifidus will be performed on MR images
Rapid reaction time | 12 weeks
  Measurement of rapid reaction time will be conducted in surface electromyo gram

CONTACTS AND LOCATIONS:
Overall Officials: maosheng Xu, Doctor, Principal Investigator — The First Affiliated Hospital of Zhejiang Chinese Medical University; honhquan Song, Bachelor, Principal Investigator — The First Affiliated Hospital of Zhejiang Chinese Medical University; hui Wei, Bachelor, Principal Investigator — The First Affiliated Hospital of Zhejiang Chinese Medical University
Locations (1):
- The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tsuji T, Matsuyama Y, Sato K, Hasegawa Y, Yimin Y, Iwata H. Epidemiology of low back pain in the elderly: correlation with lumbar lordosis. J Orthop Sci. 2001;6(4):307-11. doi: 10.1007/s007760100023. PMID 11479757